CLINICAL TRIAL: NCT05221164
Title: 162 mg of Aspirin for Prevention of Preeclampsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Methodist Medical Center of Illinois (Other)
Collaborators: University of Illinois College of Medicine at Peoria (Other); UICOM Peoria Family Medicine Residency (Unknown)
Responsible Party: Principal Investigator, Paul M Goldsmith, DO, Resident Physician, Methodist Medical Center of Illinois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1732470-3
Record Dates: First submitted 2021-08-23; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention with 162 mg aspirin (Experimental): Aspirin 162 mg daily for prevention of preeclampsia in pregnant patients at Family Medicine Clinic
  Interventions: Drug: Aspirin 162 mg

INTERVENTIONS:
Drug: Aspirin 162 mg — Daily aspirin 162 mg during pregnancy to prevent preeclampsia
  Other Names: Aspirin

SUMMARY:
This is a study to assess if 162 mg of aspirin will decrease rates of preeclampsia in pregnant patients compared to 81 mg of aspirin.

DETAILED DESCRIPTION:
After screening to meet inclusion criteria, pregnant patients at the Family Medicine Clinic will be asked to take 162 mg aspirin daily for 6 months, starting at about 12 weeks gestation and continued until the end of pregnancy. They will be monitored every 4 weeks until week 28, then every 2 weeks until week 36, and then weekly from week 36 on. Participants will be screened at these visits for medication compliance (taking, missed doses, side effects, etc). Patients will be subject to lab work as is routinely indicated for preeclampsia.

At the end of the study period, accumulated study data will be compared with historical data from the Family Medicine Clinic on rates of preeclampsia and outcomes in patients taking 81 mg for preeclampsia prevention.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant patient at Peoria FMC
* Hx of pre-eclampsia
* Multifetal gestation
* Chronic hypertension
* Type 1 or 2 diabetes
* Autoimmune disease
* Renal disease
* Nulliparity
* Obesity
* Family Hx of pre-eclampsia
* Sociodemographic characteristics
* Age >= 35 years of age
* Personal history factors (LBW, SGA, > 10-year pregnancy interval, adverse pregnancy outcomes

Exclusion Criteria:

* At high risk of side effects from ASA therapy
* Hx of hemorrhagic stroke
* Hx of GI bleed, G6PD
* Liver disease
* NSAID or Salicylate allergy)
* Patients confirmed to be not compliant with therapy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-06-09 (Estimated); Study Completion 2022-06-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with preeclampsia | Through study completion, estimated 18 months
  Dangerous pregnancy complication characterized by high blood pressure
Number of participants with eclampsia | Anytime during pregnancy and 3 months post partum
  new onset of seizures in pregnant woman with preeclampsia

SECONDARY OUTCOMES:
Number of participants with placental abruption | Through study completion, estimated 18 months
  Separation of placenta from the uterus prior to delivery
Number of participants with post partum hemorrhage | Through study completion, estimated 18 months
  blood loss after delivery
Number of participants with aplastic anemia | Through study completion, estimated 18 months
  deficiency of all blood cell lines
Number of participants with agranulocytosis | Through study completion, estimated 18 months
  deficiency of granulocytes
Number of participants with anaphylaxis | Through study completion, estimated 18 months
  serious allergic reaction

CONTACTS AND LOCATIONS:
Locations (1):
- UnityPoint Clinic Family Medicine, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD for statistical analysis and study report.
Supporting Information: SAP, CSR
Time Frame: After study completion for analysis and completion of final publication.
Access Criteria: Statistician access.

REFERENCES:
- [Result] ACOG Committee Opinion No. 743: Low-Dose Aspirin Use During Pregnancy. Obstet Gynecol. 2018 Jul;132(1):e44-e52. doi: 10.1097/AOG.0000000000002708. PMID 29939940
- [Result] Rolnik DL, Wright D, Poon LCY, Syngelaki A, O'Gorman N, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Nicolaides KH. ASPRE trial: performance of screening for preterm pre-eclampsia. Ultrasound Obstet Gynecol. 2017 Oct;50(4):492-495. doi: 10.1002/uog.18816. Epub 2017 Aug 24. PMID 28741785
- [Result] Atallah A, Lecarpentier E, Goffinet F, Doret-Dion M, Gaucherand P, Tsatsaris V. Aspirin for Prevention of Preeclampsia. Drugs. 2017 Nov;77(17):1819-1831. doi: 10.1007/s40265-017-0823-0. PMID 29039130
- [Result] Duley L, Meher S, Hunter KE, Seidler AL, Askie LM. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2019 Oct 30;2019(10):CD004659. doi: 10.1002/14651858.CD004659.pub3. PMID 31684684
- [Result] Kumar N, Das V, Agarwal A, Pandey A, Agrawal S, Singh A. Pilot Interventional Study Comparing Fetomaternal Outcomes of 150 mg Versus 75 mg Aspirin Starting Between 11 and 14 Weeks of Pregnancy in Patients with High Risk of Preeclampsia: A Randomized Control Trial. J Obstet Gynaecol India. 2020 Feb;70(1):23-29. doi: 10.1007/s13224-019-01277-5. Epub 2019 Sep 20. PMID 32030002
- [Result] Levy G. Clinical pharmacokinetics of aspirin. Pediatrics. 1978 Nov;62(5 Pt 2 Suppl):867-72. PMID 724339
- [Result] Needs CJ, Brooks PM. Clinical pharmacokinetics of the salicylates. Clin Pharmacokinet. 1985 Mar-Apr;10(2):164-77. doi: 10.2165/00003088-198510020-00004. PMID 3888490
- [Result] Roberge S, Nicolaides K, Demers S, Hyett J, Chaillet N, Bujold E. The role of aspirin dose on the prevention of preeclampsia and fetal growth restriction: systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Feb;216(2):110-120.e6. doi: 10.1016/j.ajog.2016.09.076. Epub 2016 Sep 15. PMID 27640943
- [Result] Rolnik DL, Nicolaides KH, Poon LC. Prevention of preeclampsia with aspirin. Am J Obstet Gynecol. 2022 Feb;226(2S):S1108-S1119. doi: 10.1016/j.ajog.2020.08.045. Epub 2020 Aug 21. PMID 32835720
- [Result] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Result] Seidler AL, Askie L, Ray JG. Optimal aspirin dosing for preeclampsia prevention. Am J Obstet Gynecol. 2018 Jul;219(1):117-118. doi: 10.1016/j.ajog.2018.03.018. Epub 2018 Mar 26. No abstract available. PMID 29588190